CLINICAL TRIAL: NCT07226466
Title: Evaluating Biomarkers of Cognitive Dysfunction in Patients With Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 249213; NCI-2025-01532 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumor Adult; Brain Metastases From Solid Tumors; Brain Tumor, Primary; Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Blood Specimen Collection; Quality of Life; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with Brain Tumor Receiving Radiotherapy: The study entails longitudinal assessment of plasma biomarkers (Aβ, GFAP, phospho Tau, NfL), determination of APOE genotype, neuropsychiatric testing Brain Health Assessment test (BHA), a clinically validated neurocognitive battery compiling metrics on memory and language), and brain morphometric measurements synchronized with standard of care brain MRIs.
  Interventions: Procedure: Blood sample; Procedure: Brain magnetic resonance imaging (MRI); Procedure: Brain Health Assessment; Radiation: Quality of Life (QoL) Questionnaire

INTERVENTIONS:
Procedure: Blood sample — Blood sample will be collected
Procedure: Brain magnetic resonance imaging (MRI) — Brain MRI will be performed during the course of data collection
Procedure: Brain Health Assessment — Brain Health Assessment will be performed during the course of data collection
Radiation: Quality of Life (QoL) Questionnaire — QoL questionnaire will be given to participants during the course of data collection

SUMMARY:
This study investigates the effects of brain radiotherapy on cognitive function by evaluating plasma biomarkers and apolipoprotein E (APOE) genotype in patients with primary or metastatic brain tumors. Standard brain radiotherapy is known to impact cognitive outcomes, yet the underlying biological mechanisms remain unclear.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. Assess plasma biomarkers for Aβ, GFAP, phospho Tau, and NfL pre- and post-radiotherapy.
2. Determine APOE genotype.
3. Evaluate neuropsychiatric testing aligned with standard of care brain MRIs and serum markers.
4. Measure brain morphometrics pre- and post-radiotherapy with standard of care brain MRIs.

SECONDARY OBJECTIVES:

1. Measure patient-reported quality of life changes pre- and post-radiotherapy using a standard University of California, San Francisco (UCSF) -approved questionnaire.

OUTLINE:

This is a single-arm, non-randomized, open-label pilot study. Participants will be study duration spans 12 months post-brain radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. >= 18 years old
2. Diagnosis of a primary brain tumor OR #3. Not both #2 and #3.
3. Diagnosis of primary solid tumor and secondary involvement of the brain
4. If the patient has brain metastases: fewer than 5 brain metastases (post-operative and definitive allowed), none > 1 cm in max diameter.
5. Candidate for standard of care / usual care (SOC) focused brain radiotherapy.
6. No prior brain radiotherapy, including whole brain radiotherapy.
7. Eastern Cooperative Oncology Group (ECOG) functional score 0 or 1.
8. Estimated life expectancy post-treatment of > 2 years.

Exclusion Criteria:

1. Diagnosis of neurodegenerative disease (Alzheimer's disease, Parkinson's disease).
2. Diagnosis of memory disorder pre-treatment.
3. Leptomeningeal disease or disease involving either hippocampus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with brain cancers receiving care at University of California, San Francisco (UCSF)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in serum Amyloid-beta peptide (Aβ) | Up to 12 months
  Mean change in biomarker for Aβ over time will be reported
Mean change in serum Amyloid-beta peptide (Aβ) by APOE genotype | Up to 12 months
  Mean change in biomarker for Aβ by APOE genotype over time will be reported
Mean change of score on the European Organization for Research and Treatment of Cancer quality of life questionnaire - Brain Module (EORTC-QLQ-BN20) | Up to 18 months from date of first radiation dose
  The EORTC QLQ-BN20 consists of 20 questions; seven single item symptom scales (headaches, seizures, drowsiness, hair loss, itchy skin, leg weakness and bladder control), along with four multi-item scales (future uncertainty, visual disorder, motor dysfunction and communication deficit). Raw scores for the QLQ-BN20 items are computed by calculating the mean of the items in each subscale, or the item for each individual and linearly transform the scores to a 0-100 scale. A higher score represents worse QOL for all QLQ-BN20 scales and single items.
Mean change in serum Glial Fibrillary Acidic Protein (GFAP) | Up to 12 months
  Mean change in biomarker for GFAP over time will be reported
Mean change in serum Glial Fibrillary Acidic Protein (GFAP) by APOE genotype | Up to 12 months
  Mean change in biomarker for GFAP by APOE genotype over time will be reported
Mean change in serum Phosphorylated TAU (p-TAU) | Up to 12 months
  Mean change in biomarker for p-TAU over time will be reported
Mean change in serum Phosphorylated TAU (p-TAU) by APOE genotype | Up to 12 months
  Mean change in biomarker for p-TAU by APOE genotype over time will be reported
Mean change in serum Neurofilament Light Chain (NfL) | Up to 12 months
  Mean change in biomarker for NfL over time will be reported
Mean change in serum Neurofilament Light Chain (NfL) by APOE genotype | Up to 12 months
  Mean change in biomarker for NfL by APOE genotype over time will be reported
Mean change in Brain Health Assessment by APOE genotype | Up to 12 months
  Mean change in of Brain Health Assessment by APOE genotype over time will be reported
Mean change in Hippocampal Volume | Up to 12 months
  Mean change in Hippocampal Volume as measured by MRI over time will be reported
Mean change in Hippocampal Volume by APOE genotype | Up to 12 months
  Mean change in Hippocampal Volume as measured by MRI by APOE genotype over time will be reported

SECONDARY OUTCOMES:
Change in scores on the European Organization for Research and Treatment of Cancer quality of life questionnaire 30 (EORTC-QLQ-C30) over time | Up to 18 months from date of first radiation dose
  The functional domains measure the quality of life in Physical functioning, Role functioning, Emotional functioning, Cognitive functioning, Social functioning. Scores consists of responses to items with responses ranging from 1="Not at all" to 4="Very Much". The raw score is calculated by estimating the mean of the items that make up each domains with a resulting total range of 1 - 4. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the functional domains represents a high level of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Nakamura, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No